CLINICAL TRIAL: NCT00966056
Title: Comparative Study of Mitomycin C and Internal Nasal Septal Splint in the Treatment of Nasal Synechiae
Brief Title: Study of Mitomycin C and Nasal Splint to Treat Nasal Synechiae
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karnataka Institute of Medical Sciences (Other)
Responsible Party: Dr SRINISH G, KARNATAKA INSTITUTE OF MEDICAL SCIENCES
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01_M012_3210
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2009-08

CONDITIONS: Nasal Synechiae; Adhesions of Nasal Cavity; Nasal Adhesions; Tissue Adhesions
Keywords: Nasal adhesions; Nasal synechiae; Mitomycin; Mitomycin c; Teflon; Splints; Septal splints
MeSH Terms: conditions — Tissue Adhesions | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin C (Active Comparator): Cases recruited into this arm receive topical application of mitomycin c (1mg/ml)following surgical synechiolysis
  Interventions: Drug: Mitomycin C
- Teflon septal splint (Active Comparator): Cases recruited into this arm receive insertion of teflon internal nasal septal splint following surgical synechiolysis
  Interventions: Device: Teflon nasal septal splint

INTERVENTIONS:
Drug: Mitomycin C — Cotton wick soaked with 1mg/ml of mitomycin c placed for 2 minutes between the raw surfaces after synechiolysis with surgical blade no.15
  Other Names: Mitomycin, Mitocin, MMC
  Arms: Mitomycin C
Device: Teflon nasal septal splint — Teflon internal nasal septal splint placed between the raw surfaces and secured at the anterior end of septum with catgut 3-0 sutures, following synechiolysis with surgical blade no.15. Splint removed at the end of one week
  Other Names: Teflon splint, nasal septal splint, internal nasal splint
  Arms: Teflon septal splint

SUMMARY:
This study evaluates whether Mitomycin C is an effective alternative to septal splints in the treatment of nasal synechiae.

DETAILED DESCRIPTION:
Nasal synechiae is an important cause for the failure of many a nasal surgery. Septal splints have been widely used for the treatment of nasal synechiae, but are associated significant morbidity until removal. To the best of our knowledge there are no studies in literature comparing Mitomycin C with septal splints as an atraumatic alternative in the treatment of nasal synechiae. This is a preliminary study taken up to evaluate the therapeutic efficacy of Mitomycin C in the treatment of nasal synechiae.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasal mucosal synechiae due to surgical or non-surgical trauma

Exclusion Criteria:

* Patients with nasal vestibular stenosis
* Patients with nasal synechiae due to diseases like Hansen's disease, Syphilis, Rhinoscleroma, Atrophic Rhinitis etc.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Recurrence or absence of synechiae | 1 week, 1 month, 2 months

SECONDARY OUTCOMES:
Symptoms and complications | 1 week, 1 month, 2 months

CONTACTS AND LOCATIONS:
Overall Officials: VIKRAM K BHAT, MS(ENT), DNB, Study Chair — Karnataka Institute of Medical Sciences
Locations (1):
- Karnataka Institute of Medical Sciences, Hubli, Karnataka, India